CLINICAL TRIAL: NCT04494165
Title: The Effects of Massage With Frankincense and Myrrh Oil in Treating Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Massage With Frankincense and Myrrh Oil in Treating Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ülkü özdemir, assistant professor doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019/460
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Low Back Pain
Keywords: Massage; Low Back Pain; Aromatherapy; Chronic Pain; Activities of Daily Living
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Massage; Frankincense; Carrier State

STUDY DESIGN:
Intervention Model Description: 3x2 (experiment, control and placebo group x pre-test post-test) split plot design
Who Masked: Participant, Outcomes Assessor
Masking Description: The measurements and evaluations of the patients were conducted by an independent surveyor (assessor-blind) to ensure that the study was double-blind. Massage application, the main intervention of the study, was carried out by another nurse who was trained on this subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy Group (Experimental): In addition to the standard physical therapy session, 30 patients in this group received a total of six sessions of lumbar massage for three weeks with frankincense and myrrh essential oils, two sessions per week (2nd and 5th days of each week), each lasting 15 minutes. During the massage, an average of 3ml mixture prepared by adding 2% frankincense oil and 2% myrrh essential oil to jojoba carrier oil was used as an oil mixture.
  Interventions: Other: massage with frankincense and myyrh essential oil
- placebo group (Placebo Comparator): In addition to the standard physical therapy session, 31 patients in this group received a total of six sessions of lumbar massage for three weeks with jojoba oil, two sessions per week (2nd and 5th days of each week), each lasting 15 minutes.
  Interventions: Other: massage with carrier oil
- control group (No Intervention): 30 patients in this group received standard physical therapy sessions, and no massage was applied.

INTERVENTIONS:
Other: massage with frankincense and myyrh essential oil — In addition to the standard physical therapy session, 30 patients in aromatherapy group received a total of six sessions of lumbar massage for three weeks with frankincense and myrrh essential oils, two sessions per week (2nd and 5th days of each week), each lasting 15 minutes. During the massage, an average of 3ml mixture prepared by adding 2% frankincense oil and 2% myrrh essential oil to jojoba carrier oil was used as an oil mixture.
  Arms: Aromatherapy Group
Other: massage with carrier oil — In addition to the standard physical therapy session, 31 patients in placebo group received a total of six sessions of lumbar massage for three weeks with jojoba oil, two sessions per week (2nd and 5th days of each week), each lasting 15 minutes.
  Arms: placebo group

SUMMARY:
This randomized controlled study was conducted to determine the effect of massage with frankincense and myrrh oil in treating chronic low back pain.

A total of 91 individuals over the age of 18 who agreed to participate in the study, who had no verbal communication problems, and who had complaints of low back pain for at least the past three months were included in the study. In this research, 3x2 (experiment, control and plasebo group x pre-test post-test) split plot design was used The data were collected using the data sheet, Visual Analogue Scale (VAS), Aberdeen Low Back Pain Scale (ALBPS) and Roland-Morris Disability Scale (RMDS). Standard treatment was applied to all three groups for three weeks, every weekday. In addition to the standard treatment, 2 sessions of waist massage per week were applied to the aromatherapy Group with frankincense and myyrh essential oil and to the Placebo Group with jojoba fixed oil in accordance with the aromatherapy protocol. Massage was not applied to the control group.

In the results of working, the decrease in RMDS (p <0.001), ALBPS (p <0.001) and VAS (p <0.001) scores of the aromatherapy group was found to be statistically higher than the other two groups.

As a result, aromatherapy massage with Fankincense and Myyrh essential oil can be added to traditional treatments as an easy-to-apply complementary health application with no significant side effects to relieve pain and reduce disability in an individual's daily life in chronic low back pain patient care.

DETAILED DESCRIPTION:
The research was conducted as a randomized, double-blinded, placebo-controlled study to examine the effect of massage with frankincense and myrrh essential oils on pain and disability in individuals with chronic low back pain. In this research, 3x2 (experiment, control and placebo group x pre-test post-test) split plot design was used. The measurements and evaluations of the patients were conducted by an independent surveyor (assessor-blind) to ensure that the study was double-blind. Massage application, the main intervention of the study, was carried out by another nurse who was trained on this subject.

Individuals presenting with chronic low back pain, who were admitted to the physical medicine and rehabilitation outpatient clinic of a training and research hospital and who were prescribed a physical therapy session constituted the target population of the study.

For the sample size, 30-31-30 patients were included in the experimental, placebo and control groups, between June and October 2019, respectively, and power analysis was performed with the obtained data. As a result of power analysis, the effect size for Roland-Morris Disability Scale (RMDS) was 0.44 and statistical power was 100%; the effect size for Aberdeen Low Back Pain Scale (ALBPS) was 0.53 and the statistical power was 100%; and the effect size for Visual Analogue Scale (VAS) was 0.29 and statistical power was 100%, and the research was completed.

Individuals who meet the inclusion criteria were included in the randomization pool and then assigned to one of the following groups:

1. Aromatherapy Group which had classical massage with essential oil,
2. Placebo Group which had classical massage with a fixed oil,
3. Control Group. Pre-application was made to 5 individuals to check the functionality of the forms and application. In the pre-application, it was decided that only effleurage and friction should be performed, since the individuals were disturbed by petrissage during massage. After pre-application, the study was finalized. Individuals who participated in pre-application were not included in the study.

Informed consent of the individuals randomly assigned to the groups was obtained. There was no intervention in the standard treatment applied in the clinic. At the beginning of the study, VAS, ALBPS, RMDS were applied to all three groups prior to the intervention by face-to-face interview method. Then, all three groups received standard treatment for three weeks, every weekday. In addition to the standard treatment, aromatherapy group was applied 2 sessions of 15 min lumbar massage per week (2nd and 5th day) with frankincense and myrrh essential oils, and the placebo group was applied lumbar massage with jojoba fixed oil in the same frequency. Massage was not applied to the control group. After three weeks, VAS, ALBPS, RMDS were applied to all 3 groups after the intervention Massage Application: Although there are many massage techniques, the most widely used technique is Swedish massage technique applied with light pressure. Swedish massage is a superficial massage and has a stimulating effect on soft tissues and blood circulation. The main maneuvers of classical massage are effleurage, petrissage, friction, tapotement and vibration. In this study, effleurage and friction were applied from these maneuvers.

Effleurage is a stroking movement applied on the skin with one hand or both hands. In the stroking technique, palms, fingers, thumb and back of hand is applied with one or two hands. The aim is to accelerate blood flow in superficial veins and excretion of metabolites from the body. Friction is the pressing, scrubbing and sliding movements with small circular movements using fingertips, thumbs, four fingers and palms. The purpose of friction is to remove adhesions in skin and subcutaneous tissue, to relax stiffness and thickening, to reduce fluid in tissues around joints and to remove metabolites.

Essential oils from plants are used topically for massaging, often by adding them into carrier oil The use of essential oils in massage is called aromatherapy massage. In this study, frankincense and myrrh essential oils were used as essential oil and jojoba oil was used as carrier oil.

Intervention: The standard physical therapy session of the clinic lasts for three weeks (3x5=15 sessions in total, 30 minutes on average per session) on a weekday basis. During the session, hot pack, ultrasound therapy and TENS (trans electrical nerve stimulation) were applied. The lumbar massage performed as a research intervention was performed immediately after the physical therapy session to increase the effectiveness of the intervention.

Intervention applied to the aromatherapy group: In addition to the standard physical therapy session, 30 patients in this group received a total of six sessions of lumbar massage for three weeks with frankincense and myrrh essential oils, two sessions per week (2nd and 5th days of each week), each lasting 15 minutes. During the massage, an average of 3ml mixture prepared by adding 2% frankincense oil and 2% myrrh essential oil to jojoba carrier oil was used as an oil mixture.

Intervention applied to the placebo group: In addition to the standard physical therapy session, 31 patients in this group received a total of six sessions of lumbar massage for three weeks with jojoba oil, two sessions per week (2nd and 5th days of each week), each lasting 15 minutes.

Intervention applied to the control group: 30 patients in this group received standard physical therapy sessions, and no massage was applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18,
* who agreed to participate in the study,
* who had no communication problems (hearing, vision, speech, perception problem)
* who had been suffering from (chronic) low back pain for at least the past three months were included in the study.

Exclusion Criteria:

* Patients with allergic skin reactions,
* those who had undergone a surgical operation or fracture in the lumbar region in the last year,
* those with a fever above 38.5 °C,
* those undergoing a neurological rehabilitation,
* patients with active infections such as tuberculosis and AIDS,
* those undergoing cancer treatment,
* those who had received massage therapy for the last three months were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | three weeks
  It is stated that VAS is more sensitive and reliable than other one-dimensional scales in the measurement of pain intensity(*). In their study, Cline, Herman, Show et al. (1992) have reported that vertical use of VAS is better understood by patients. (*). It was used in our study to assess the severity of low back pain. It is a-10 cm ruler with endpoints of "no pain" at one end and "unbearable pain" at the other end. The scale was explained to the patient and they were asked to mark any place between these two points that matched the severity of their pain. The distance between the beginning of "no pain" and the point marked by the patient was measured and recorded in centimeters.
Aberdeen Low Back Pain Scale | three weeks
  It is a scale that patients can fill out by themselves to decide on the health status of patients with low back pain. It is a 19-item scale consisting of questions about number of days with pain, use of painkillers, factors that increase and decrease pain, pain areas, sensory change, loss of strength/weakness, lumbar flexion, difficulty falling asleep due to pain, sitting, getting up, walking, work/daily activities, sex life, leisure activities, self-care, and days spent in bed. The total score of the scale adapted to Turkish by İlhanlı et al. ranges between 0 and 100, and the high score indicates more severe low back pain. Its Cronbach's Alpha value was indicated as 0.88 (*). In our study, the power of the scale was 100%.
Roland-Morris Disability Scale | three weeks
  The patient is asked to mark the appropriate ones among the 24 cases specified in this form. RMDS consists of 24 expressions based on the patient's perception of low back pain and associated disability. These items are indicated as physical activity (15), sleep/rest (3), psychosocial (2), household management (2), eating (1) and frequency of pain (1) (*).This test is based on measuring how low back pain affects the patient's activities of daily living. Yes responses are calculated as "1", no responses as "0" points, and a total score between 0 and 24 is obtained. Higher score means more disability. The Turkish validity study of the scale was conducted by Küçükdeveci et al. Cronbach's alpha value of the scale was indicated as 0.85-0.89 (*). In our study, the power of the scale was 100%

CONTACTS AND LOCATIONS:
Overall Officials: ülkü özdemir, Principal Investigator — erciyes üniversitesi
Locations (1):
- Ülkü Özdemir, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no planing

REFERENCES:
- [Derived] Alkanat HO, Ozdemir U, Kulakli F. The effects of massage with frankincense and myrrh oil in chronic low back pain: A three-arm randomised controlled trial. Explore (NY). 2023 Sep-Oct;19(5):761-767. doi: 10.1016/j.explore.2023.04.004. Epub 2023 Apr 14. PMID 37121835